CLINICAL TRIAL: NCT06696248
Title: The Efficacy of Carvedilol Combined with Compound Alverine Citrate Soft Capsules in the Treatment of Portal Hypertension in Patients with Liver Cirrhosis: a Prospective, Open-label, Multicentre, Randomised Controlled Trial
Brief Title: Carvedilol and Alverine in Portal Hypertension
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shanghai East Hospital (Other); Army Medical Center of PLA (Other Government)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-PH-ALV-2403
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hypertension, Portal
Keywords: Cirrhotic portal hypertension; Alverine; Pharmacological therapy
MeSH Terms: conditions — Hypertension, Portal | interventions — Carvedilol; alverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carvedilol + Alverine Group (Experimental): On the basis of maintaining unchanged routine hepatoprotective and symptomatic supportive treatments and the original dose of carvedilol, participants will be administered with compound alverine citrate capsules (Le Jian Su; specification: each capsule contains alverine citrate 60 mg and simeticone 300 mg; manufactured by Laboratoires MAYOLY SPINDLER), at a dosage of 180 mg/day (1 capsule orally, 3 times a day), for a continuous period of 24 weeks.
  Interventions: Drug: Carvedilol and alverine

INTERVENTIONS:
Drug: Carvedilol and alverine — On the basis of maintaining unchanged routine hepatoprotective and symptomatic supportive treatments and the original dose of carvedilol, participants will be administered with compound alverine citrate capsules (Le Jian Su; specification: each capsule contains alverine citrate 60 mg and simeticone 300 mg; manufactured by Laboratoires MAYOLY SPINDLER), at a dosage of 180 mg/day (1 capsule orally, 3 times a day), for a continuous period of 24 weeks.

SUMMARY:
Brief summaries of CZXH-PH-ALV-2403 The goal of this clinical trial is to learn if the combination of alverine and carvedilol works to treat portal hypertension in adult patients with liver cirrhosis. It will also learn about the safety of alverine.

The main question it aims to answer is:

For patients with liver cirrhosis and portal hypertension who have been treated with carvedilol at a dose of up to 15 mg/day or at a lower dose that is the maximum tolerated for at least 3 months, and still have a hepatic venous pressure gradient (HVPG) of 12 mmHg or higher and up to and including 20 mmHg, can the addition of alverine help to reduce portal hypertension? On the basis of maintaining unchanged routine hepatoprotective and symptomatic supportive treatments and the original dose of carvedilol, participants will be administered with compound alverine citrate capsules (Le Jian Su; specification: each capsule contains alverine citrate 60 mg and simeticone 300 mg; manufactured by Laboratoires MAYOLY SPINDLER), at a dosage of 180 mg/day (1 capsule orally, 3 times a day), for a continuous period of 24 weeks.

DETAILED DESCRIPTION:
1. Study Overall Design This trial is a prospective, single-arm, multicenter, exploratory clinical trial. Subjects who meet the inclusion criteria and do not meet the exclusion criteria enter a 24-week treatment period after signing the informed consent form. In addition to the baseline period, subjects undergo efficacy assessment 24 weeks after treatment. The safety of carvedilol combined with alverine treatment for portal hypertension in patients with liver cirrhosis is evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0; safety is assessed through laboratory tests, 12-lead electrocardiograms, and vital signs, physical examinations, etc.
2. Study Purpose 2.1 Primary Study Purpose To evaluate the efficacy of carvedilol combined with compound alverine citrate capsules in the treatment of portal hypertension in patients with liver cirrhosis.

   2.2 Secondary Study Purposes 2.2.1 To evaluate the effect of carvedilol combined with compound alverine citrate capsules on the incidence of esophageal and gastric variceal bleeding and other decompensating events in cirrhosis; 2.2.2 To evaluate the safety of carvedilol combined with compound alverine citrate capsules in the treatment of portal hypertension in patients with liver cirrhosis.
3. Study Endpoints 3.1 Primary Endpoint The proportion of patients who achieve a reduction in HVPG of ≥10% from baseline or a reduction to below 12mmHg after 24 weeks of treatment (the treatment response rate).

   3.2 Secondary Endpoints 3.2.1 The reduction in HVPG from baseline levels after 24 weeks of treatment; 3.2.2 The incidence of decompensating events in cirrhosis during the treatment period (esophageal and gastric variceal bleeding and rebleeding, new-onset ascites/progression of ascites, spontaneous bacterial peritonitis, overt hepatic encephalopathy, acute kidney injury/hepatorenal syndrome, etc.); 3.2.3 The treatment response rate at 12 weeks; 3.2.4 The reduction in HVPG from baseline HVPG after 12 weeks of treatment; 3.2.5 The reduction in mean arterial pressure of subjects after treatment compared to baseline values; 3.2.6 The reduction in heart rate of subjects after treatment compared to baseline values; 3.2.7 The incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment (evaluated according to CTCAE version 5.0).
4. Study Population 4.1 Inclusion Criteria 4.1.1 Ages 18 to 80 years old (inclusive), no gender restrictions; 4.1.2 Patients with liver cirrhosis diagnosed by clinical, laboratory, imaging examinations, and/or liver biopsy; 4.1.3 Treated with carvedilol at a dose of up to 15 mg/day or at a lower dose that is the maximum tolerated for at least 3 months, with HVPG≥12 mmHg and ≤20 mmHg; 4.1.4 Agree to participate and sign the informed consent form. 4.2 Exclusion Criteria 4.2.1 Those who have taken alverine, papaverine, or their derivatives (such as papaverine hydrochloride preparations, trimebutine maleate, etc.) within 4 weeks before enrollment; 4.2.2 Those who have undergone transjugular intrahepatic portosystemic shunt (TIPS) or other interventional treatments affecting portal pressure (including splenic embolization, splenic microwave treatment, etc.) or liver transplantation; 4.2.3 Those who have had overt hepatic encephalopathy, esophageal and gastric variceal bleeding within 2 weeks before enrollment; those who have undergone endoscopic treatment for esophageal and gastric varices within 1 week before enrollment or are planned for endoscopic treatment; 4.2.4 Those who have used somatostatin and its analogs, vasopressin, terlipressin, dopamine, norepinephrine, and other vasoactive drugs within 1 week before enrollment; 4.2.5 Those with a history of heavy alcohol consumption within 12 weeks before enrollment and cannot abstain from alcohol during the study period (equivalent ethanol intake of ≥30 g/day for males and ≥20 g/day for females); 4.2.6 Serum total bilirubin levels ≥3×ULN (for patients with autoimmune liver disease, serum total bilirubin levels ≥5×ULN), or serum sodium levels <125 mmol/L, or white blood cell count <1×10^9/L, or platelet count <30×10^9/L, or International Normalized Ratio (INR) >1.8; or serum creatinine ≥1.2×ULN; 4.2.7 Presence of thrombosis in the portal venous system (including portal vein, splenic vein, superior mesenteric vein, etc.) and cavernous transformation of the portal vein; those with a history of portal venous system thrombosis who have no definite thrombosis detected in the portal venous system within 2 weeks before enrollment may be included; 4.2.8 HBV DNA or HCV RNA > the lower limit of detection; patients with active hepatitis C receiving antiviral treatment; those who have received anti-HBV treatment for less than 24 weeks; 4.2.9 Those with uncontrollable current infections (pulmonary infections, abdominal infections, HIV, etc.) within 4 weeks before enrollment; 4.2.10 Those with poorly controlled hypertension, diabetes, or other severe heart, lung diseases; 4.2.11 Those diagnosed or suspected to have malignant tumors, including liver cancer; 4.2.12 Known allergies to alverine, papaverine, or their derivatives (such as papaverine hydrochloride preparations, trimebutine maleate, etc.), or simethicone, or carvedilol; patients with contraindications to carvedilol: New York Heart Association Class IV decompensated heart failure requiring intravenous inotropic agents; asthma, chronic obstructive pulmonary disease (COPD) with bronchospasm; second- or third-degree atrioventricular block, severe bradycardia (heart rate less than 50 beats per minute), sick sinus syndrome (including sinoatrial block); cardiogenic shock; severe hypotension (systolic blood pressure less than 85 mmHg); 4.2.13 Those with glaucoma; 4.2.14 Those with mental abnormalities; 4.2.15 Pregnant or breastfeeding women, or women who do not rule out the possibility of pregnancy; 4.2.16 Those who have participated in other drug trials within 4 weeks before enrollment; 4.2.17 Other reasons the investigator deems unsuitable for participation.
5. Intervention On the basis of maintaining unchanged routine hepatoprotective and symptomatic supportive treatments and the original dose of carvedilol, participants will be administered with compound alverine citrate capsules (Le Jian Su; specification: each capsule contains alverine citrate 60 mg and simeticone 300 mg; manufactured by Laboratoires MAYOLY SPINDLER), at a dosage of 180 mg/day (1 capsule orally, 3 times a day), for a continuous period of 24 weeks.
6. Sample size calculation This exploratory clinical trial plans to include 30 participants.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 80 years old (inclusive), no gender restrictions;
* Patients with liver cirrhosis diagnosed by clinical, laboratory, imaging examinations, and/or liver biopsy;
* Treated with carvedilol at a dose of up to 15 mg/day or at a lower dose that is the maximum tolerated for at least 3 months, with HVPG≥12 mmHg and ≤20 mmHg;
* Agree to participate and sign the informed consent form.

Exclusion Criteria:

* Those who have taken alverine, papaverine, or their derivatives (such as papaverine hydrochloride preparations, trimebutine maleate, etc.) within 4 weeks before enrollment;
* Those who have undergone transjugular intrahepatic portosystemic shunt (TIPS) or other interventional treatments affecting portal pressure (including splenic embolization, splenic microwave treatment, etc.) or liver transplantation;
* Those who have had overt hepatic encephalopathy, esophageal and gastric variceal bleeding within 2 weeks before enrollment; those who have undergone endoscopic treatment for esophageal and gastric varices within 1 week before enrollment or are planned for endoscopic treatment;
* Those who have used somatostatin and its analogs, vasopressin, terlipressin, dopamine, norepinephrine, and other vasoactive drugs within 1 week before enrollment;
* Those with a history of heavy alcohol consumption within 12 weeks before enrollment and cannot abstain from alcohol during the study period (equivalent ethanol intake of ≥30 g/day for males and ≥20 g/day for females);
* Serum total bilirubin levels ≥3×ULN (for patients with autoimmune liver disease, serum total bilirubin levels ≥5×ULN), or serum sodium levels <125 mmol/L, or white blood cell count <1×10^9/L, or platelet count <30×10^9/L, or International Normalized Ratio (INR) >1.8; or serum creatinine ≥1.2×ULN;
* Presence of thrombosis in the portal venous system (including portal vein, splenic vein, superior mesenteric vein, etc.) and cavernous transformation of the portal vein; those with a history of portal venous system thrombosis who have no definite thrombosis detected in the portal venous system within 2 weeks before enrollment may be included;
* HBV DNA or HCV RNA > the lower limit of detection; patients with active hepatitis C receiving antiviral treatment; those who have received anti-HBV treatment for less than 24 weeks;
* Those with uncontrollable current infections (pulmonary infections, abdominal infections, HIV, etc.) within 4 weeks before enrollment;
* Those with poorly controlled hypertension, diabetes, or other severe heart, lung diseases;
* Those diagnosed or suspected to have malignant tumors, including liver cancer;
* Known allergies to alverine, papaverine, or their derivatives (such as papaverine hydrochloride preparations, trimebutine maleate, etc.), or simethicone, or carvedilol; patients with contraindications to carvedilol: New York Heart Association Class IV decompensated heart failure requiring intravenous inotropic agents; asthma, chronic obstructive pulmonary disease (COPD) with bronchospasm; second- or third-degree atrioventricular block, severe bradycardia (heart rate less than 50 beats per minute), sick sinus syndrome (including sinoatrial block); cardiogenic shock; severe hypotension (systolic blood pressure less than 85 mmHg);
* Those with glaucoma;
* Those with mental abnormalities;
* Pregnant or breastfeeding women, or women who do not rule out the possibility of pregnancy;
* Those who have participated in other drug trials within 4 weeks before enrollment;
* Other reasons the investigator deems unsuitable for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The 24-week response rate | 24 weeks
  The response rate to treatment, defined as the percentage of patients with a decrease in HVPG of ≥10% from baseline or a decrease to below 12 mmHg after 24 weeks of treatment.

SECONDARY OUTCOMES:
Degree of decrease in HVPG compared to baseline HVPG after 24 weeks of treatment. | 24 weeks
Incidence of cirrhosis decompensation events during treatment. | 24 weeks
  Incidence of cirrhosis decompensation events (including esophageal and gastric variceal bleeding, new-onset ascites/progression of ascites, spontaneous bacterial peritonitis, overt hepatic encephalopathy, acute kidney injury/hepatorenal syndrome, primary liver cancer, etc.) during treatment.
The 12-week response rate | 12 weeks
  The response rate to treatment, defined as the percentage of patients with a decrease in HVPG of ≥10% from baseline or a decrease to below 12 mmHg after 12 weeks of treatment.
Degree of decrease in HVPG compared to baseline HVPG after 12 weeks of treatment. | 12 weeks
Degree of decrease in mean arterial pressure (MAP) compared to baseline MAP after 24 weeks of treatment. | 24 weeks
Degree of decrease in heart rate (HR) compared to baseline HR after 24 weeks of treatment. | 24 weeks
Incidence of Treatment-Emergent Adverse Events [Safety assessment] | 24 weeks
  The incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment The incidence of adverse events, serious adverse events, and adverse events leading to treatment discontinuation after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, M.D., Principal Investigator — Shanghai Changzheng Hospital